CLINICAL TRIAL: NCT00693784
Title: A Multicenter Pilot Study of Resorbable Biologic Disc Augmentation for Treatment of Symptomatic Lumbar Internal Disc Disruption (IDD) With the Biostat® Disc Augmentation System
Brief Title: Treatment of Symptomatic Lumbar Internal Disc Disruption (IDD) With the Biostat® Disc Augmentation System: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spinal Restoration, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SR-BX01P-2007
Record Dates: First submitted 2008-06-04; First posted 2008-06-09 (Estimated); Results first posted 2010-04-29 (Estimated); Last update posted 2015-06-22 (Estimated); Status verified 2015-05

CONDITIONS: Low Back Pain
Keywords: Intervertebral Disk; chronic low back pain; internal disc disruption; degenerative disc disease
MeSH Terms: conditions — Low Back Pain; Intervertebral Disc Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Biostat® Disc Augmentation System (Experimental): Delivery of Biostat BIOLOGX® Fibrin Sealant with the Biostat Delivery Device
  Interventions: Biological: Biostat® Disc Augmentation System

INTERVENTIONS:
Biological: Biostat® Disc Augmentation System — Delivery of Biostat BIOLOGX® Fibrin Sealant with the Biostat Delivery Device

SUMMARY:
The purpose of this study is to assess the safety of the Biostat Disc Augmentation System for the treatment of chronic low-back (lumbar) pain due to symptomatic internal disc disruptions (IDD) and to obtain preliminary efficacy information.

DETAILED DESCRIPTION:
The Biostat Disc Augmentation System is a combination product combining a resorbable biologic product with a delivery device system used to prepare and insert the biologic material into a lumbar intervertebral disc.

Symptomatic IDD is defined as a painful disruption of the internal architecture of a lumbar intervertebral disc, which appears as fissures, cracks or tears within the internal structures of the disc. Pain arising from a lumbar disc may not only be perceived as pain located in the low back (axial pain), but also as somatic referred pain involving the posterior hips, buttock, lateral hips, groin, or posterior thighs.

The diagnosis of symptomatic IDD cannot currently be made on the basis of imaging studies, physical examination, or symptoms alone, and must be established with meticulously conducted disc provocation studies (provocation discography) that include pressure manometry, and identification of an adjacent normal disc.

This treatment and study are not designed for patients exhibiting other potential sources of chronic low back pain such as more advanced degenerative disc disease with significant loss of disc height (> 33%), spinal stenosis, or spondylolisthesis (see Eligibility Criteria).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 (inclusive) and skeletally mature.
* Voluntarily signs the subject informed consent form and agrees to the release of medical information for purposes of this study (HIPAA authorization).
* Physically and mentally able to comply with the protocol, including ability to read and complete required forms, and willing and able to adhere to the follow-up requirements of the protocol.
* Low-back pain for at least 6 months.
* Pretreatment baseline low-back pain of at least 40 mm on a 100 mm visual analog scale.
* Referred leg pain, if present, is of noncompressive origin and there are no clinical findings of radiculopathy.
* Low-back pain is greater than leg pain (if present) as measured on a visual analog scale. If bilateral leg pain, back pain is greater than worst leg pain.
* Low-back pain unresponsive to at least 6 weeks of nonoperative treatment, which may include bed rest, antiinflammatory and analgesic medications, chiropractic manipulations, acupuncture, massage, physical therapy or home-directed lumbar exercise program.
* Negative response to diagnostic medial branch block or facet joint injection.
* No sustained relief with epidural injection of corticosteroids.
* Diagnosis of symptomatic lumbar (L1/L2-L5/S1) internal disc disruption (IDD), which requires confirmation of discogenic pain at one or two contiguous levels through positive provocation discography performed using pressure manometry and identification of an adjacent normal disc. The disc provocation studies must precisely demonstrate concordant pain (<50 psi above opening pressure) and must demonstrate a fissure(s) in the outer one-third of the posterior or lateral anulus.

Exclusion Criteria:

* Cauda equina syndrome.
* Active malignancy or tumor as source of symptoms.
* Infection at the planned procedure site or active systemic infection.
* Previous lumbar spine surgery.
* Previous disc invasive treatment procedures at the affected level(s) (e.g., intradiscal electrothermal therapy, intradiscal radiofrequency thermocoagulation) in the past 12 months or intradiscal corticosteroid injection within the past 3 months.
* Evidence of prior lumbar vertebral body fracture or trauma.
* Disc bulge/protrusion at the symptomatic level(s) > 4 mm.
* Presence of disc extrusion or sequestration.
* Clinical findings of lumbosacral motor or sensory radiculopathy.
* Leg pain is greater than low-back pain as measured on a visual analog scale.
* Lumbar intervertebral foramen stenosis at the affected level(s) resulting in significant spinal nerve root compression or impingement.
* Symptomatic central vertebral canal stenosis or absolute sagittal vertebral canal diameter < 9mm.
* Loss of disc space height at the symptomatic level(s) greater than one-third of an adjacent normal disc (or of the expected height in the case of an L5-S1 disc).
* Spondylolisthesis (≥ Grade 1) with or without spondylolysis at the symptomatic level(s).
* Lumbar spondylitis or other undifferentiated spondyloarthropathy.
* Dynamic instability on lumbar flexion-extension radiographs.
* Positive response to diagnostic medial branch block or facet joint injection.
* Positive response to diagnostic sacroiliac joint injection for those patients with pain in the sacral region
* Sustained relief obtained with epidural injection of corticosteroids.
* Symptomatic involvement of more than two lumbar disc levels.
* Congenital or acquired coagulopathy or thrombocytopenia; or currently taking anticoagulant, antineoplastic, antiplatelet, or thrombocytopenia-inducing medications.
* History of unexplained, easy, or persistent bruising or bleeding, bleeding from the gums, or bleeding problems experienced in previous surgical procedures.
* Aspirin or aspirin-containing medication taken ≤7 days prior to the procedure.
* Significant systemic disease, including unstable angina, autoimmune disease, rheumatoid arthritis, and muscular dystrophy.
* Known or suspected hypersensitivity or allergy to drugs or components of the fibrin sealant, including aprotinin, used in the procedure.
* History of, or current psychiatric condition, substance or alcohol abuse that would potentially interfere with the subject's participation in the study.
* Ongoing or previous participation in another drug or device clinical study within the previous 2 months.
* Subject known to be pregnant or nursing at time of enrollment or with plans to become pregnant within the planned length of follow-up (2 years).
* Body habitus precludes adequate fluoroscopic visualization for the procedure or the procedure is physically impossible using the device.
* Concomitant conditions requiring daily oral steroid usage for more than 30 days in the preceding 90 days.
* Pending litigation against a health care professional, except where required by the insurer as a condition of coverage.
* Prisoner or active military personnel who would not be available for follow-up.
* Presence of ferromagnetic implants that would disallow MRI of the symptomatic disc(s).
* Active or pending workers' compensation claims.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-06; Primary Completion 2009-02 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin J Pauza, MD, Principal Investigator — Spine Specialists, PA
Locations (3):
- United States (3):
  - Bethesda, Maryland
  - Tyler, Texas
  - Bellingham, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- BIOSTAT BIOLOGX: 1 injection of from 1 to 4 mL of BIOSTAT BIOLOGX Fibrin Sealant
Period: Overall Study
Arm/Group | BIOSTAT BIOLOGX
Started | 15
26-Week Primary Endpoint | 15
52-week Extended Follow-up | 13
104-week Extended Follow-up | 11
Completed | 11
Not Completed | 4
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | BIOSTAT BIOLOGX
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 13
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.9 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Numbers and Types of Adverse Events (Only Number of Events is Reported in This Section - See Adverse Events Section for Further Detail)
Description: The primary outcome for this safety study includes the number and types of adverse events reported in the study. The data fields in this section do not allow for reporting all aspects of this outcome (i.e., the number of adverse events, as well as the types of event). These numbers were entered and are reported in the adverse event section of the Results.
Time Frame: 104 weeks
Population: All 15 participants available through 26-week primary endpoint. One voluntary withdrawal and 1 lost-to-follow-up between 26-week follow-up and 52-week extended follow-up. One additional voluntary withdrawal and 1 additional lost-to-follow-up between 52-week extended follow-up and 104-week extended follow-up.
Measure: Number; unit: Events
Arm/Group | BIOSTAT BIOLOGX
Number analyzed (Participants) | 15
Events | 17

2. Secondary Outcome: Visual Analog Scale for Low-back Pain
Description: 100 mm line anchored on the left with the descriptor "No pain" (best value = 0 mm) and anchored on the right with the descriptor "Worst possible pain" (worst value = 100 mm). Lower scores indicate less pain.
Time Frame: Baseline, 26-weeks (primary endpoint), 52-weeks, 104-weeks
Population: n=15 (all participants at baseline and 26-week primary endpoint) n=13 at 52 weeks n=11 at 104 weeks
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | BIOSTAT BIOLOGX
Number analyzed (Participants) | 15
mm
  Baseline | 72.4 (14.2)
  26-wks | 31.7 (26.0)
  52-wks | 35.4 (29.3)
  104-wks | 33.0 (24.8)

3. Secondary Outcome: Roland-Morris Disability Questionnaire
Description: 24-item questionnaire with score determined by the number of items checked by the subject. Items assess the effect of back pain on limitations of normal daily activities. Best value = 0 (least disability). Worst value = 24 (most disability). Higher number indicate greater disability.
Time Frame: Baseline, 26-weeks (primary endpoint), 52-weeks, 104-weeks
Population: n=15 (all participants at baseline and 26-week primary endpoint) n=13 at 52 weeks n=11 at 104 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | BIOSTAT BIOLOGX
Number analyzed (Participants) | 15
Units on a scale
  Baseline | 15.2 (4.5)
  26-weeks | 8.9 (6.5)
  52-weeks | 6.2 (4.7)
  104-weeks | 5.6 (4.1)

ADVERSE EVENTS:
Time Frame: 104 weeks
Arm/Group | BIOSTAT BIOLOGX
Serious Adverse Events (participants affected / at risk) | 2/15
Other Adverse Events (participants affected / at risk) | 9/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIOSTAT BIOLOGX (N=15)
Discitis (Infections and infestations) | 1 (1)
Tumor (Renal and urinary disorders) | 1 (1) — Kidney tumor present but undetected at baseline.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIOSTAT BIOLOGX (N=15)
Muscle spasm (Musculoskeletal and connective tissue disorders) | 2 (2)
Buttock Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Herpes (Immune system disorders) | 1 (1)
Trip/fall (General disorders) | 3 (3)
Motor vehicle accident (General disorders) | 1 (2)
Low back pain (Musculoskeletal and connective tissue disorders) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days